CLINICAL TRIAL: NCT00440323
Title: A Double-blind, Double-dummy, Randomised, Placebo-controlled,Four-way Crossover Study to Investigate the Effect of Single Oral Doses of SB-649868 and of Zolpidem in a Model of Noise Induced Situational Insomnia in Healthy Male Volunteers.
Brief Title: Disturbed Sleep Model Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: OXS104094
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Noise induced Situational insomnia,; healthy volunteers; SB-649868,; Zolpidem,
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — N-((1-((5-(4-fluorophenyl)-2-methyl-4-thiazolyl)carbonyl)-2-piperidinyl)methyl)-4-benzofurancarboxamide; Zolpidem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ADBC sequence (Experimental): In ADBC sequence A is Placebo, B is SB-649868 10 milligram (mg), C is SB-649868 30 mg, and D is Zolpidem 10 mg. Subject will receive placebo tablets, then two 5 mg tablets of SB-649868, then 25 mg and 5 mg tablet of SB-649868. There will be wash-out period of 7 days.
  Interventions: Drug: SB-649868; Drug: Zolpidem; Drug: Placebo
- BACD sequence (Experimental): In BACD sequence subject will receive SB-649868 two tablets of 5 mg each (10 mg, B), Placebo tablets (A), SB-649868 two tablets of 25 mg and 5 mg (30 mg, C), and Zolpidem 10 mg (D). There will be wash-out period of 7 days.
  Interventions: Drug: SB-649868; Drug: Zolpidem; Drug: Placebo
- CBDA sequence (Experimental): In CBDA sequence subject will receive SB-649868 two tablets of 25 mg and 5 mg (30 mg, C), SB-649868 two tablets of 5 mg each (10 mg, B), Zolpidem 10 mg (D) and Placebo tablet (A). There will be wash-out period of 7 days.
  Interventions: Drug: SB-649868; Drug: Zolpidem; Drug: Placebo
- DCAB sequence (Experimental): In DCAB sequence subject will receive Zolpidem 10 mg (D), SB-649868 two tablets of 25 mg and 5 mg (30 mg, C), Placebo tablet (A), and SB-649868 two tablets of 5 mg each (10 mg, B). There will be wash-out period of 7 days.
  Interventions: Drug: SB-649868; Drug: Zolpidem; Drug: Placebo

INTERVENTIONS:
Drug: SB-649868 — SB-649868 tablets will be available with dose strength of 5 and 25 mg.
Drug: Zolpidem — Zolpidem capsules will be available with dose strength of 10 mg.
  Other Names: SB-649868
Drug: Placebo — Placebo tablet matching SB-649868 or Placebo capsule matching Zolpidem will be available.

SUMMARY:
Subjects will be screened within 28 days. Each treatment session will consist of 2 PSG nights, study drug administration and noise model is conducted on second night.

ELIGIBILITY:
Inclusion Criteria:

* Body weight =50 kg and BMI within the range 18.5-29.9 kg/m2 inclusive
* Healthy as judged by responsible physician.
* No clinically significant abnormality identified on the medical or laboratory evaluation and 12-lead ECG;
* The subject shows a normal sleep pattern on the basis of the evaluation of both PSG screening nights. Normal sleep will be defined as follows: LPS (Latency to persistence Sleep) <30min., SE (Sleep Efficiency) >85%, apnea/ hypopnea index < 10, periodic leg movements (PLM) with arousal index < 10. The apnea/hypopnea index is defined as "the number of apneas and hyponeas divided by the total sleep time (TST) expressed in hours". PLMI is defined as "the number of periodic leg movements associated with arousals or awakening divided by the total sleep time (TST) expressed in hour".

Exclusion Criteria:

* A positive result for the pre-study urine drug/ alcohol breath screen.
* Abuse of alcohol.
* Subject complains of sleep disturbances and /or is receiving treatment for sleep disorders.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2007-01-05 (Actual); Primary Completion 2007-07-03 (Actual); Study Completion 2007-07-03 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time measured overnight across four treatment sessions (4 weeks) | 4 weeks

SECONDARY OUTCOMES:
The effects on daytime cognitive function following dosing across four treatment sessions (4 weeks) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Guildford, Surrey, United Kingdom

REFERENCES:
- [Derived] Bettica P, Squassante L, Groeger JA, Gennery B, Winsky-Sommerer R, Dijk DJ. Differential effects of a dual orexin receptor antagonist (SB-649868) and zolpidem on sleep initiation and consolidation, SWS, REM sleep, and EEG power spectra in a model of situational insomnia. Neuropsychopharmacology. 2012 Apr;37(5):1224-33. doi: 10.1038/npp.2011.310. Epub 2012 Jan 11. PMID 22237311
- See also: Results for study OXS104094 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/OXS104094?search=study&search_terms=OXS104094#rs